CLINICAL TRIAL: NCT06983652
Title: Validation of the Use of Terahertz Scanning System on Corneal Scars and Corneal Edema: Phase II Clinical Trial
Brief Title: Validation of the Use of Terahertz Scanning System on Corneal Scars and Corneal Edema
Status: Recruiting | Type: Observational
Sponsor: Singapore Eye Research Institute (Other)
Responsible Party: Sponsor
Other Study IDs: 2024-3286
Record Dates: First submitted 2025-05-06; First posted 2025-05-21 (Actual); Last update posted 2025-05-21 (Actual); Status verified 2025-05

CONDITIONS: Corneal Diseases; Corneal Scars and Opacities; Corneal Edema
Keywords: cornea; corneal scar; corneal edema; Terahertz; hydration
MeSH Terms: conditions — Corneal Diseases; Corneal Injuries; Corneal Edema

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Corneal edema cohort: Patients with corneal endothelial dysfunction (Fuchs' endothelial dystrophy or other causes of bullous keratopathy) at any disease stage, with manifestation of corneal edema.
  Interventions: Device: THz scanning using THz Imaging system.
- Corneal scar cohort: Patients with corneal scars from any cause, with the absence of corneal edema.
  Interventions: Device: THz scanning using THz Imaging system.

INTERVENTIONS:
Device: THz scanning using THz Imaging system. — The THz scanning system is non-invasive and non-contact. It is a prototype developed by Institute of Materials Research and Engineering (IMRE), A*STAR, Singapore and is performed for the purpose of research. THz scanning will provide safety data in human and the measurement of cornea hydration status. Each THz scan will take approximately 1 second. Real-time data will be generated when participants are positioned in front of the device.

SUMMARY:
This observational study aims to validate the use of THz scanning system in corneal edema and corneal scars, and to investigate the accuracy and performance on the use of THz scanning system in the evaluation of the progression of corneal edema and corneal scars. Participants corneal scars and corneal edema will undergo THz scanning, followed by a series of conventional clinical examinations for detailed characterization of the corneal lesion. The performance of the use of THz system on corneal scars and edema will be evaluated by correlating measurements from the THz scans with those obtained from standard clinical methods. The investigators hypothesize that the THz scanning system has the capacity to evaluate the hydration level on human corneas.

DETAILED DESCRIPTION:
Corneal opacity is one of the main causes of low vision and visual impairment, which results from two pathological etiologies: corneal edema and corneal scarring. When corneal opacity progresses to end-stage disease, the only option is to undergo a corneal transplantation. There is a global shortage of donor corneas and patients who undergo corneal transplantation require life-long topical immunosuppressant treatment, hence monitoring the progression of corneal edema or corneal scarring to prevent the disease entering into the end stage is crucial. Monitoring the progression of diseases also allows surgeons to do earlier intervention with less invasive techniques, such as lamellar corneal graft, as opposed to full-thickness graft. Currently there is no objective tool clinically to quantitatively evaluate corneal opacity and there is no tool to directly evaluate corneal hydration level. Hence, there is a need to develop a quantitative tool to evaluate the density of corneal opacities. There is a need to develop a medical tool to evaluate the corneal scar objectively and quantitatively, to better monitor the disease progression and aid in the surgical decision making.

Terahertz (THz) waves are electromagnetic radiation, and have emerged as a novel, non-invasive and non-contact imaging modality in the biomedical field, with a fast-scanning speed (30ms per scan) to meet medical diagnostic needs. With its fast scanning, it provides a more accurate result for the estimation of corneal thickness. Its high sensitivity hydration absorption and characterization peaks of collagen will provide a useful tool to obtain information that are related to the corneal layers. Water has a high dielectric constant and is highly absorptive to THz spectrum. This allows THz wave to be highly sensitive to water content in tissue. Furthermore, THz scan has been applied to a variety of hydration-related diseases or conditions. With THz scan, early detection of disease and diagnosis can be carried out. Some examples would be the prediction of skin flap failure, diagnosis for the presence of caries lesion at its initial stage, identification of skin cancer in skin biopsy samples and to access the physiological dynamics of tear film in dry eye syndrome. Previous studies have demonstrated that THz scanning system could be used as an early diagnostic tool, to identify the cancerous area based on the lack of clear cellular order in the skin. It was able to detect disease conditions in deeper layers, allowing it to be an effective early diagnostic tool for basal cell carcinoma. Moreover, it had been confirmed that THz scanning system had the sensitivity to identify the difference in colon tissue composition. The findings showed that the properties of ex vivo tissue, had an increase in both absorption coefficient and refractive indices in disease tissue when compared to healthy tissue. A recent study showed that with THz scanning system, clinicians will be able to obtain different images, such as 3D imaging methods to provide multiple views of internal structures. Furthermore, with the THz scan, the process of water loss in an in vitro porcine corneal tissue could be determined using a THz reflection imaging system. It was found that THz wave was approximately linear to the water content concentration, and that the slope decreased monotonously with an increase in frequency. Thus THz imaging is suggested to be used for the clinical diagnosis of corneal edema or scars, dry eye diseases and corneal hydration in refractive surgery.

The investigators would like to conduct the clinical trial to validate the use of THz scanning system in human corneal edema and corneal scars.

ELIGIBILITY:
Inclusion Criteria:

* Be at least 21 years of age.
* Regardless of gender (Male/Female).
* Regardless of race (Chinese/Malay/Indian/Eurasian/Others).
* Willingness and ability to follow all instructions and comply with study schedule for study visit.
* Patients with corneal endothelial dysfunction (Fuchs' endothelial dystrophy or other causes of bullous keratopathy) at any disease stage OR Patients with corneal scars from any cause, with the absence of corneal edema.
* Ability to hold face sufficiently stable to undergo necessary scans.

Exclusion Criteria:

* Eyes with active inflammation or infection, or chronic ocular surface inflammation
* Unable to give consent
* Physically immobile/poor instructional compliance
* PI determined
* Pregnant/ breast feeding women

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A total of 150 participants with corneal diseases, including corneal scars and corneal edema, will be recruited from Singapore National Eye Centre.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2024-07-01 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
National Eye Institute (NEI) Score | Baseline
  The cornea will be divided into five regions, each scored ranging from 0 (no fluorescein staining) to 3 (severe fluorescein staining) according to the grading scheme. The total NEI score will range from 0 to 15.
Central corneal thickness | Baseline
  Central corneal thickness (CCT) will be assessed using Anterior Segment Optical Coherence Tomography. The CCT will be measured using a build-in caliper software.
Measurements of corneal scars | Baseline
  Segment Optical Coherence Tomography will be used to perform 1x corneal cross line scan, and 3x 3D cornea scans to obtain detailed measurements of the corneal scars. All scans will be taken en-face.
Level of corneal density | Baseline
  Corneal densitometry will be performed using the rotating Scheimpflug anterior segment analyzer. All parameters will be automatically calculated by the in-built software and densitometry measurements will be expressed in standardized greyscale units.
Extent of keratocytes activation | Baseline
  In vivo confocal microscopy will be used to capture images of keratocytes. The gray values of reflectivity for corneal stromal scans will be semi-quantified to confirm if there are significant changes in the activity of stromal keratocytes.
Overall appearance of corneas | Baseline
  External eye photos will be captured to record the status of corneas, showing the location and extent of involvement of the corneal lesion.

CONTACTS AND LOCATIONS:
Locations (1):
- Singapore National Eye Centre, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No